CLINICAL TRIAL: NCT02866695
Title: Safety and Efficacy of Ingenol Mebutate Gel 0.015% for Treatment of Actinic Keratosis on the Face in Solid Organ Transplant Recipients
Brief Title: Safety and Efficacy of Ingenol Mebutate Gel 0.015% for Treatment of AK on the Face in Solid Organ Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Leo AK
Record Dates: First submitted 2016-08-02; First posted 2016-08-15 (Estimated); Results first posted 2019-02-25 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Actinic Keratosis
Keywords: Actinic Keratosis; lung transplant; kidney transplant
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label treatment (Other): All patients will be treated with ingenol mebutate gel 0.015%. There is no placebo or comparator for this study. The investigator will identify the patient's treatment area at Baseline, and provide a detailed application instruction sheet. The first dose will be applied in clinic under the supervision of the investigator.
  Interventions: Drug: ingenol mebutate gel 0.015%

INTERVENTIONS:
Drug: ingenol mebutate gel 0.015% — ingenol mebutate gel 0.015% to be applied on treatment area
  Other Names: Picato

SUMMARY:
This is a single arm, open-label interventional study of ingenol mebutate 0.015% in solid organ transplant recipients. The investigators plan to treat 20 subjects, 10 kidney transplant recipients and 10 lung transplant recipients. The investigators have selected these two populations as the represent the spectrum of solid organ transplantation: kidney transplant recipients are the largest transplant population, but have lower levels of immunosuppression and skin cancer risk. Lung transplant recipients have the highest burden of skin cancer and actinic keratoses.

DETAILED DESCRIPTION:
Actinic keratoses (AK) are patches of dysplastic keratinocytes arising in sun-damaged skin. These lesions are precursors to cutaneous squamous cell carcinoma (SCC), and are treated to prevent progression to SCC. First-line therapy for AK include cryotherapy and curettage, which target clinically visible lesions but do not address the subclinical lesions in the field of ultraviolet radiation damage. Field therapy includes topical chemotherapy, immunotherapy, and photodynamic therapy. Ingenol mebutate is the active compound found in Euphorbia peplus sap, and has been approved for treatment of AK in immunocompetent patients. Ingenol mebutate 0.015% is favored over other topical treatments for treatment of AK on the face due to the brief treatment course, high clearance rate, and resolution without sequelae.

Solid organ transplant recipients (OTR) have a high incidence of AK and high risk of developing SCC, and require frequent field therapy. In addition, OTR generally have a higher burden of AK and require treatment of a larger surface area than the 25 cm2 area labeled for ingenol mebutate 0.015%. The investigators plan to investigate the safety and efficacy of ingenol mebutate 0.015% in OTR, with a treatment area up to 100cm2.

This is a single arm, open-label interventional study of ingenol mebutate 0.015% in solid organ transplant recipients. The investigators plan to treat 20 subjects, 10 kidney transplant recipients and 10 lung transplant recipients. The investigators have selected these two populations as the represent the spectrum of solid organ transplantation: kidney transplant recipients are the largest transplant population, but have lower levels of immunosuppression and skin cancer risk. Lung transplant recipients have the highest burden of skin cancer and actinic keratoses.

ELIGIBILITY:
Inclusion Criteria:

1. Adults at least 18 years old.
2. Subject must be a solid organ transplant recipient at least one year from the date of transplantation.
3. Subjects must be in stable health as confirmed by medical history, per investigator judgement.
4. Subjects must be able to read, sign, and understand the informed consent.
5. Subjects have at least 4 and no more than 20 clinically typical (non-hyperkeratotic/hypertrophic), visible actinic keratoses in a treatment area of approximately 100cm2 on the face. Treatment areas will include a single cheek (nasofacial sulcus to tragus, malar cheekbone to jawline and avoiding the lower eyelid and mouth); the forehead (hairline to eyebrows, extending laterally to the root of the helix).
6. Subject must be willing to forego any other treatments on the face, including cryotherapy, tanning bed use and excessive sun exposure while in the study.
7. Subject is willing and able to participate in the study and to comply with all study requirements including concomitant medication and other treatment restrictions.
8. If subject is a female of childbearing potential she must have a negative urine pregnancy test result prior to study treatment initiation and must agree to use an approved method of birth control while enrolled in the study.

Exclusion Criteria:

1. Subjects with an unstable medical condition as deemed by the clinical investigator.
2. Subjects with a history of bone marrow or stem cell transplantation.
3. Subjects with non-melanoma skin cancer on the face.
4. Subjects with hyperkeratotic or hypertrophic AKs.
5. Subjects with any dermatologic disease in the treatment area that may be exacerbated by the treatment proposed or that might impair the evaluation of AKs.
6. Women who are pregnant, lactating, or planning to become pregnant during the study period.
7. Subjects who have previously been treated with ingenol mebutate in study area within the past 8 weeks.
8. Subjects who have used any topical prescription medications for actinic keratosis on the study area within 8 weeks prior to study treatment initiation.
9. Subjects who have used any topical prescription medications for other reason on the study area within 4 weeks prior to study treatment initiation.
10. Subjects who are currently participating in another clinical study or have completed another clinical study with an investigational drug or device on the study area within 30 days prior to study treatment initiation.
11. Subjects with known hypersensitivity to Picato gel or any of the inactive ingredients: isopropyl alcohol, hydroxyethyl cellulose, citric acid monohydrate, sodium citrate, or benzyl alcohol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Arron, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Dermatology, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be shared with authorized representatives of the study sponsor LEO Pharma, Inc., The University of California, FDA

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label Treatment: A total of 20 solid organ transplant recipients with 4 to 20 actinic keratoses were enrolled and treated for 3 consecutive days with 4 single-dose tubes of ingenol mebutate gel 0.015% applied to a 100 cm2 area of the face according to study protocol. There was no placebo or comparator for this study. All but 2 participants completed the treatment. One kidney transplant participant forgot to apply the treatment on day 3, but continued in the study. One lung transplant participant who reported pain in the treatment area withdrew from the study after day 2 dosing due to travel considerations and was lost to follow-up.
Period: Overall Study
Arm/Group | Open Label Treatment
Started | 20
Completed | 18
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Treatment
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 65.3 [42.1 to 75.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
Organ Transplant Type [Count of Participants; unit: Participants]
  Lung | 9
  Kidney | 7
  Kidney/Pancreas | 2
  Kidney/Liver | 1
  Kidney/Heart | 1
Years Since Transplant [Mean (Full Range); unit: years] | 10.9 [1 to 33]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: To evaluate the safety of ingenol mebutate gel 0.015% on the face in solid organ transplant recipients
Time Frame: From screening to Day 57 or study early termination if applicable
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Treatment
Number analyzed (Participants) | 20
Participants
  Facial edema | 12
  Pain in Treatment Area | 11
  Pruritus | 6
  Headache | 3
  Squamous Cell Carcinoma Outside Treatment Area | 3
  Diarrhea | 2
  Xerosis | 2
  Urosepsis | 1
  Worsening of CKD | 3
  Hyperglycemia | 2
  Acute Kidney Injury | 1
  Hyperkalemia | 1
  Anemia | 1
  Hypertriglyceridemia | 1

2. Secondary Outcome: Number of Participants With a Reduction of Actinic Keratosis
Description: To evaluate the efficacy of ingenol mebutate for reduction of actinic keratoses on the face in organ transplant recipients.
Time Frame: Day 57 (assessed at screening, day 1, day 29, day 57, and study early termination if applicable, clearance at day 57 reported)
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Treatment
Number analyzed (Participants) | 20
Participants
  75% Clearance of Actinic Keratoses at Day 57 | 12
  100% Clearance of Actinic Keratoses at Day 57 | 8

3. Secondary Outcome: Participant's Local Skin Response Grading Scale
Description: To investigate the local skin response to ingenol mebutate in organ transplant recipients. Local skin reaction (LSR) will be graded by visual assessment on a 4 point scale where 0=none, 1=mild, 2=moderate, 3=severe. Each of the following four reactions will be graded: erythema, vesiculation/postulation, crusting/scabbing/erosion, and edema/swelling. A composite score will be calculated (range 0-16). A high LSR indicated a worse outcome. LSR assessment will be performed at days 1, 8, 29, and 84.
Time Frame: Day 1, Day 4 (assessed at screening, day 1, day 4, day 29, day 57, and study early termination if applicable, results at day 1 and day 4 reported)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label Treatment
Number analyzed (Participants) | 20
score on a scale
  Baseline Local Skin Reaction Composite Score | 1.2 (0.8)
  Day 4 Local Skin Reaction Composite Score | 11.7 (4.2)

ADVERSE EVENTS:
Time Frame: Each participant was assessed for 57 days from the start of treatment.
Description: CTC Adverse Events Grading Criteria version 4.0 was used to define adverse events
Arm/Group | Open Label Treatment
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 5/20
Other Adverse Events (participants affected / at risk) | 10/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Treatment (N=20)
Urosepsis (Renal and urinary disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Chronic Kidney Disease (Renal and urinary disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Treatment (N=20)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Acute Kidney Injury (Renal and urinary disorders) | 4 (4)
Hyperkalemia (Renal and urinary disorders) | 1 (1)
Hypocalcemia (Renal and urinary disorders) | 1 (1)
Hyponatremia (Renal and urinary disorders) | 2 (2)
Hypoalbuminemia (Renal and urinary disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-18): https://cdn.clinicaltrials.gov/large-docs/95/NCT02866695/Prot_SAP_000.pdf